CLINICAL TRIAL: NCT02627859
Title: A 26 Week Multicenter Prospective Open Label Clinical Study Evaluating a Single Intra-articular Injection of DUROLANE SJ1ml for Treatment of OA Pain of the Ankle
Brief Title: 26 Week Open Label Study Evaluating Single IA Injection of DUROLANE SJ for Treatment of Osteoarthritis Pain of the Ankle
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bioventus LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13DUR502
Record Dates: First submitted 2015-12-08; First posted 2015-12-11 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Durolane SJ (Experimental): Durolane SJ intra-articular injection; device
  Interventions: Device: Durolane SJ

INTERVENTIONS:
Device: Durolane SJ — 1ml single intra-articular injection in ankle

SUMMARY:
26 week open label study of treatment with Durolane for OA pain of the ankle

DETAILED DESCRIPTION:
Single injection Durolane in patients with mild to moderate OA of the ankle.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males between the ages of 19 and 85 years of age
2. Diagnosis of mild to moderate (K-L grade II or III) osteoarthritis (OA) of the study ankle joint, confirmed by radiographs taken within the previous six months OA in the contralateral ankle is permissible provided that OA symptoms are greater in the study ankle.
3. VAS (100mm) AOS pain subscale score in the range of 30mm to 90mm for the study ankle
4. Must be willing to discontinue use of oral and topical analgesia other than rescue use of acetaminophen for any pain including OA pain in the study ankle. Must also be willing to discontinue acetaminophen rescue medication for at least 24 hours before each study visit
5. Abstinence from any IA or peri-articular injections in the study ankle during the course of the trial, except for the Investigational Product
6. Cooperative and able to communicate effectively with the Investigators
7. Patients with chronic ankle pain of the study ankle lasting more than 6 months without clinically significant improvement in ankle pain over the past one month
8. Body mass index (BMI) ≤ 35 kg/m2.
9. English literacy and ability to understand and complete all informed consent procedures

Exclusion Criteria:

1. Significant pain from other joints or low back pain requiring chronic ongoing analgesic therapy
2. Hindfoot deformities
3. Substantial venous or lymphatic stasis in the legs
4. Presence of one or more conditions that could confound pain and functional assessments in the study ankle, e.g., plantar fasciitis, Achilles tendonitis, sprains of the foot, or degenerative joint disease of the foot.
5. Clinically-apparent tense effusion, signs of misalignment or instability in the study ankle
6. Ankle x-ray findings of acute fractures, severe loss of bone density, avascular necrosis and/or severe deformity in the study ankle
7. Surgery to the study ankle within the previous 12 months
8. Unable to abstain treatment with NSAIDs or any pain management medications during the week (or five half-lives of the drug, whichever is longer) prior to Baseline Visit.
9. Unable to abstain from treatment with topical analgesics during the washout period prior to screening visit and throughout the duration of the study. Washout period for topical analgesics is based on clinical investigator judgment (~ a few days).
10. Inability to tolerate acetaminophen for rescue medication use.
11. IA or local peri-articular corticosteroid injections to the study ankle within the previous three months; or to any other joint within the previous month; or any oral corticosteroid within the previous month. Steroid inhalants are permitted if the patient has been on a stable regimen for the past month and remains on this regimen throughout the course of the trial
12. IA injections with hyaluronic acid in the study ankle within the last 9 months
13. Previous allergic reaction to a HA or lidocaine product allergies.
14. Treatment with glucosamine/chondroitin sulfate initiated within the past three months, or dosage not stable for the past three months
15. Change in physical therapy for the study ankle within one month preceding screening, or expected change in physical therapy for the ankle during the study
16. Planned surgical procedure during the study period.
17. Previous history or presence of septic arthritis in study ankle
18. Active skin disease or infection in the area of the injection site
19. Alcohol or drug abuse as determined by the Investigator or use of alcohol for control of pain; Use of illicit drugs including cannabis.
20. Systemic inflammatory condition or autoimmune disease or infection such as rheumatoid arthritis, inflammatory arthritis, ankylosing spondylitis, psoriatic arthritis, reactive arthritis, gout/ acute pseudo gout or any other connective tissue disease
21. Uncontrolled hypothyroidism
22. Treatment with anticoagulant (except for acetylsalicylic acid maximum of 325mg/day)
23. Any medical condition which in the opinion of the investigator makes the patient unsuitable for inclusion (e.g., severe progressive chronic disease, malignancy, bleeding disorder, fibromyalgia)
24. Pregnant or breast-feeding woman or woman of child-bearing potential not practicing adequate contraception.
25. Subjects that in the opinion of the investigator are unsuitable for inclusion (e.g., subjects not likely to avoid other therapies, subjects not likely to stay in the study or with plans to relocate during the whole study period, or subjects likely to be unreliable)
26. Concurrent participation in any other clinical study or participation within the preceding 30 days

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-06; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
AOS pain subscale score | at 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Younger, MD, Principal Investigator — St. Pauls Hospital
Locations (1):
- Providence Health Care, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes